CLINICAL TRIAL: NCT03270241
Title: Early Molecular Changes in Vitiligo After Narrowband Ultraviolet Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00133884
Record Dates: First submitted 2017-08-28; First posted 2017-09-01 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Vitiligo; Dermatology/Skin - Other
Keywords: Vitiligo; Dermatology; Johns Hopkins; Compensation; Paid; Phototherapy; NB-UVB; Light treatment; Skin; Biopsies; Money; Short-term
MeSH Terms: conditions — Vitiligo | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: Participants diagnosed with Vitiligo who are enrolled in the study will receive phototherapy (NB-UVB), with the starting dose of 250 mJ/cm2. The dose will be increased by 10% with each treatment. Small skin samples will be collected before and after NB-UVB treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Phototherapy (NB-UVB) (Experimental): Phototherapy (NB-UVB) will be administered for all enrolled subjects. The starting dosage will be 250 mJ/cm2. The dose will be increased by 10% with each treatment, as long as there are no side effects with treatment.
  Interventions: Device: Phototherapy (NB-UVB) via the 3 Series PC & SP phototherapy cabinet

INTERVENTIONS:
Device: Phototherapy (NB-UVB) via the 3 Series PC & SP phototherapy cabinet — This is an investigator-initiated, single-blinded, ascending dose study of NB-UVB treatment for Vitiligo in adults of 3 treatments for one week. It is designed to measure the molecular changes and re-pigmentation in affected and normal skin of participants with Vitiligo and normal skin in healthy participants.

SUMMARY:
Vitiligo is a chronic acquired cutaneous disease of pigmentation that affects patients' quality of life across all degrees of involvement and severity. Phototherapy, such as Narrow band UVB (NB-UVB), is a clinically indicated treatment for skin lesions. NB-UVB treatment has been shown to promote repigmentation and normalize cellular behaviors. The investigators would like to analyze the change in protein expression and histological change in skin from NB-UVB treatment in participants with Vitiligo.

The investigators are recruiting participants with Vitiligo on the body, arms, and/or legs.

DETAILED DESCRIPTION:
This is a dermatology study of the effects of short-term NB-UVB treatment, standard phototherapy for Vitiligo patients. In the study, demographics information, three ascending dose of phototherapy, and small skin biopsies will be required of the participants.

For all enrolled participants, the starting dose of NB-UVB administered will be 250 mJ/cm2, which is the standard of care for patients with Vitiligo. The dose will be increased by 10% with each treatment, as long as there are no side effects with treatment such as burning or redness/ erythema. Small skin biopsies will be collected from normal skin and from affected skin from vitiligo participants at the baseline visit and 3 days after the conclusion of treatment; up to a total of 6 biopsies will be collected from each patient. Participants will be compensated for time and effort.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older with bilateral symmetrical vitiligo lesions, in general good health as determined by the Principal Investigator by medical history and physical exam.
* Able to understand consent procedure
* Able to comply with protocol activities

Exclusion Criteria:

* Patients less than 18 years old
* Patients not able to understand consent procedure
* Patients unable to comply with protocol activities
* Non-English speakers: the study assessments/questionnaires/evaluations are not scientifically validated in languages other than English.
* Patients with a photosensitive disorder or on a medication which has been demonstrated in these patients to cause photosensitivity
* Patients receiving concomitant phototherapy to test sites
* Patient receiving topical medication to test sites within 2 weeks of study initiation
* Patient receiving oral medications for vitiligo within 4 weeks prior to study initiation
* Receipt of an investigation agent within the past 4 weeks (or within 5 half lives) prior to study initiation
* Pregnant or nursing patients (self-reported)
* Patient with significant medical history or concurrent illness that the investigator feels is not safe for study participation, including melanoma
* Presence or suspicion of bleeding disorder or diathesis which would complicate biopsy.
* Patients with history of excessive scar or keloid formation in the past 10 years
* Patients with known allergy to anesthetic used
* Subjects with a pacemaker, implanted cardioverter-defibrillator, baroreflex activation device, cochlear implant, implanted bone growth stimulator, robotic limb prosthesis, subcutaneous GPS tracking device, electrodes implanted in the brain, attached electrodes in a subject undergoing cardiac defibrillation during the moment of skin color reading, or other device which may be disrupted by electrical current, UNLESS subject is kept "1 yard (one arm's length) from the main unit" of the spectrophotometer at all times, as specified in device approval letter.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noori Kim, M.D, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Outpatient Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are still deciding on what information to release to other researchers.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phototherapy (NB-UVB)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phototherapy (NB-UVB)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 4
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Molecular Changes From NB-UVB Therapy
Description: The investigators are assessing the histological and molecular changes of normal and Vitiligo-lesion skin from NB-UVB therapy. The molecular markers (in microgram/ mL) include, but not limited to, KIT receptor, stem cell factor (SCF), tumor necrosis factor-alpha (TNF-alpha), and interleukin-1 (IL-1).
Time Frame: 2 years
Population: Data was not collected.
Arm/Group | Phototherapy (NB-UVB)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Phototherapy (NB-UVB)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phototherapy (NB-UVB) (N=10)
Wound Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT03270241/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT03270241/ICF_001.pdf